CLINICAL TRIAL: NCT01169220
Title: Single Blind, Randomized, Controlled Trial of Conventional Versus Split-Dose Bowel Preparation for Inpatient Colonoscopy
Brief Title: Bowel Preparation for Inpatient Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Santa Clara Valley Health & Hospital System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 10-041
Record Dates: First submitted 2010-07-20; First posted 2010-07-26 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Gastrointestinal Hemorrhage; Colon Cancer; Diverticulosis
Keywords: Colonoscopy; Bowel preparation
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Colonic Neoplasms; Diverticulum

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Split prep (Experimental)
  Interventions: Drug: Go Lytely
- Whole prep (Active Comparator)
  Interventions: Drug: Go-Lytely

INTERVENTIONS:
Drug: Go-Lytely — Bowel cleansing agent
  Arms: Whole prep
Drug: Go Lytely — Bowel cleansing agent
  Arms: Split prep

SUMMARY:
This study will compare two strategies for bowel cleansing prior to inpatient colonoscopy: the entire preparation taken the night before the procedure versus half the preparation taken the night before the procedure, and the other half taken the morning of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* any diagnosis for which colonoscopy is indicated

Exclusion Criteria:

* ileus
* severe colitis/toxic megacolon
* gastric retention
* bowel perforation
* gastrointestinal obstruction
* gastroparesis that precludes oral bowel preparation
* pregnant or lactating women
* allergy to polyethylene glycol.
* unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Quality of colon cleansing | 24 hours from study enrollment

SECONDARY OUTCOMES:
Patient satisfaction | 24 hours from study enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Clara Valley Medical Center, San Jose, California, United States